CLINICAL TRIAL: NCT03484169
Title: Effects of Pelvic Patterns of Proprioceptive Neuromuscular Facilitation in the Pelvic Floor Muscles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Josepha Karinne de Oliveira Ferro, PhD student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PNF in pelvic floor muscles
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Motor Activity
Keywords: Muscle Stretching Exercises; Pelvic Floor; motor control; motor skill; motor activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Will be part of the study 30 healthy women at menacme, eutrophic, nulliparous and aged between 18 and 35 years, recruited among students of the Department of Physical Therapy of the Federal University of Pernambuco. The initial sample will be divided into two groups: intervention group n=15 (GI) and one control group n=15 (CG), randomized through www.randomization.com by a researcher who will be blind regarding outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The result of the randomization will be placed in sealed and opaque envelopes and the information will be revealed to the member in charge of the training only at the moment the intervention is performed, guaranteeing the secrecy of the allocation. The study will be triple blind, since the randomization and allocation of participants will be performed by researcher A, electromyographic evaluations, data tabulation and statistical analysis (researcher B) and intervention (researcher C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention
- intervention group (Experimental): The training of PNF pelvic patterns for motor learning in GI will be performed twice a week by a trained and experienced researcher for six weeks (CHRISTIANSEN et al., 2017). At each training session, there will be three repeated movements in each pelvic pattern:
  Combination of isotonic (concentric, stabilizing and eccentric) of the anterior elevation pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the previous depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior elevation pattern;
  Interventions: Other: intervention group

INTERVENTIONS:
Other: intervention group — The training of PNF pelvic patterns for motor learning in GI will be performed twice a week by a trained and experienced researcher for six weeks (CHRISTIANSEN et al., 2017). At each training session, there will be three repeated movements in each pelvic pattern:
  Combination of isotonic (concentric, stabilizing and eccentric) of the anterior elevation pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the previous depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior elevation pattern;
  Other Names: pelvic pattern of proprioceptive neuromuscular facilitation
  Arms: intervention group

SUMMARY:
Specific patterns of PNF have been used in neurological and rheumatologic rehabilitation to improve trunk control and postural stability. However, there are no studies that analyze the effect of pelvic PNF patterns on pelvic floor muscles. We hypothesize that pelvic patterns of proprioceptive neuromuscular facilitation activate the pelvic floor muscles in healthy individuals through the abdomino-pelvic synergism. Thus, the objective of the study is to analyze the effects of pelvic patterns PNF on the recruitment of pelvic floor muscles in healthy individuals.

DETAILED DESCRIPTION:
The project will address three aspects: a) analyze the activation of the deep pelvic floor muscles during the application of pelvic PNF patterns through electromyographic measurements; b) verify which diagonals of these pelvic patterns have a better effect on the recruitment of these muscle fibers; c) to analyze electromyographic activity after motor learning (repeated training of 12 sessions).

Study Design: Randomized controlled trial.

Sample: Will be part of the study 70 healthy women at menacme, eutrophic, nulliparous and aged between 18 and 35 years, recruited among students of the Department of Physical Therapy of the Federal University of Pernambuco. The initial sample will be divided into two groups: intervention group (GI) and one control group (CG), randomized through www.randomization.com by a researcher who will be blind regarding outcomes. The result of the randomization will be placed in sealed and opaque envelopes and the information will be revealed to the member in charge of the training only at the moment the intervention is performed, guaranteeing the secrecy of the allocation. The study will be triple blind, since the randomization and allocation of participants will be performed by researcher A, electromyographic evaluations, data tabulation and statistical analysis (researcher B) and intervention (researcher C). After the initial analysis, the sample calculation will be performed using GPower software version 3.1.

Methodological outline:

Three researchers (A, B and C) will be part of the study data collection. After the clear explanation of the procedures that will be carried out during the research and the application of the Informed Consent Form (TCLE), the individuals will be subjected to a screening to analyze the eligibility. Initially, a semistructured form will be used to collect data that may be important during the analysis of the results, such as personal and sociodemographic data, anthropometric characteristics, associated diseases, medication use and gynecological history. Afterwards, the Female Sexual Function Index (FSFI) will be applied to evaluate the sexual function of the participants, translated and validated for use in Brazil.

After the application of the semistructured form, the volunteers will be submitted to a postural evaluation using photogrammetry and, physical examination for functional evaluation of the pelvic floor muscles, using the PERFECT protocol.

Finally, the electromyographic activity of the pelvic floor and abdominal muscles will be recorded during the performance of the pelvic patterns of PNF with active and resisted movements.

Recording of the electromyographic signal:

Surface electromyography will be performed during the application of pelvic PNF patterns and when associated with an active contraction of the MAP. For that, self-adhesive surface electrodes, simple and low impedance MAXICOR medical products (Paraná, Brazil), positioned in the abdominal region and pelvic floor, will be used. Owing to the rules for the acquisition of the electromyographic signal, standardized by the International Society of Electrophysiology and Kinesiology (ISEK), low-impedance surface circular electrodes (25mm diameter), self-adhesive (solid cellulose gel) and disposable surface electrodes will be used. To eliminate external interferences, a reference electrode positioned on the right anterior superior iliac spine (EIAS) will be used following the recommendations of the SENIAM (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles) Project. To minimize noise, recording and capture devices will only be connected to the battery during data collection. In order to reduce the impedance of the skin, the area will be cleaned to be positioned the electrodes using moist wipes, drying it just before registration. Also, to reduce the impedance of the skin, the tricotomy of the area where the electrode will be positioned before data collection will be requested, as well as the bladder emptying before the procedures. The electromyographic recording will be performed with the patient in left lateral decubitus during the application of pelvic PNF patterns. The general guidelines for the positioning of the electrodes described by SENIAM will be followed, however, the muscles analyzed are not included in their specific electrode placement recommendations. Therefore, to capture the electromyographic signal will be positioned along the line of action of muscle fibers, always choosing the right side of the individual, in the following anatomical structures:

* Transverse abdominal / internal oblique muscle group: surface electrode positioned 2 cm proximal to the midpoint between the pubic symphysis and the anterior superior iliac spine (EIAS).
* Lumbar square muscle: surface electrode positioned 4 cm lateral, based on the vertebral sulcus of the muscle belly of the erector muscle of the spine with slightly oblique angulation at half the distance between the 12th rib and the iliac crest.
* Thigh adductor group: upper middle third in the midline of the thigh.
* Pelvic floor muscles: in the supine position, the surface electrodes will be positioned at the three and nine o'clock position of the perineal clock.

The acquisition will be performed outside of the menstrual period and three maximal voluntary contractions (CVM) of each muscle or muscle group evaluated will be requested to obtain the highest activity during standardized tests (AEMP RMS). It will be requested the maximum contraction that the participant can perform and each contraction being sustained for 3 seconds, with interval of 30 seconds between each contraction.

After the acquisition of the AEMP RMS registry, the registry will be performed during the execution of the four isolated pelvic patterns (RMS AEMFNPI) and later when associated with pelvic floor muscle contraction (RMS AEMFNPA).

To acquire the electromyographic signal, a Miotec® surface electromyograph (Miotool 400 model, Miotec Equipamentos Biomédicos Ltd. Porto Alegre, Brazil) will be used with four channels and 14-bit analogue / digital (A / D) resolution, with internal gain of 1000 times. The sampling frequency per channel used will be 2000 Hz, 110 dB common mode rejection (CMRR), 1010 Ohm // 2pF input impedance, and fourth order Butterworth analog filter. The captured signal will be recorded using the Miotec Suite Software version 1.0 (Miotec®, Porto Alegre, Brazil) and transferred to a portable computer.

Proprioceptive Neuromuscular Facilitation Protocol:

The pelvic movements that originate the patterns are: Anterior Elevation (EA); Posterior Depression (PD); Posterior Elevation (EP) and Anterior Depression (AD) of the pelvis, totaling four specific pelvic patterns and two diagonals [anterior elevation and posterior depression (Diagonal 1) and posterior Elevation and anterior depression (Diagonal 2)] In this study, the performance of the pelvic patterns, accompanied by the electromyographic signal capture, will be performed after learning the technique done through rhythmic initiation. After learning each pattern, electromyographic recording will be performed using the specific isotonic combination technique, which combines concentric, eccentric and stabilizing contractions of the agonist muscle group without relaxation.

The protocol will be divided into four stages:

1. st stage: Initial recording of the electromyographic signal during the execution of pelvic PNF patterns.

   The electromyographic signal (RMS AEMFNPI) during the four pelvic patterns: anterior elevation, posterior elevation, anterior depression and posterior depression will be made as the lateral decubitus individual and in each muscle or muscle group evaluated during the execution of the combination technique isotonic in each pattern. The electromyographic recording of the abdominal and pelvic floor muscles will be done three times to perform the weighted average in the following sequences:

   Combination of isotonic (concentric, stabilizing and eccentric) of the anterior elevation pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior depression pattern ; Combination of isotonic (concentric, stabilizing and eccentric) of the previous depression pattern ; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior elevation pattern ;
2. nd stage: Electromyographic evaluation during a maximal voluntary contraction of each muscle or muscle group evaluated.

Participants will undergo a preparatory training to awareness of the correct contraction of the pelvic floor muscles with the guidance of a pelvic physiotherapist and later electromyographic recording (AEMP RMS) during a maximal voluntary contraction of the pelvic floor muscles as well as of the abdominal muscles, adductors of the thigh and lumbar square through the standardized tests. In order to reduce the activity of the accessory musculature during the capture of the electromyographic signal of the MAP, the individual will adopt dorsal decubitus posture with flexion and external hip rotation and knee flexion, simulating the frog posture of the Global Posture Reeducation (RPG) technique.

Stage 3: Intervention - Motor skills training The training of the pelvic PNF patterns for motor learning in the GI will be performed twice a week by a trained and experienced researcher for six weeks. At each training session, there will be three repeated movements in each pelvic pattern.

4th stage: Re-evaluation of electromyographic activity after intervention. In this stage, an electromyographic reassessment of the two groups (GI and GC) after the training period will be performed, following the same sequences of step 1 (isolated recording during the execution of the pelvic standards) and step 3 (recording during the execution of the associated pelvic patterns to the voluntary contraction of MAPs.

ELIGIBILITY:
Inclusion Criteria:

* female individuals
* aged between 18 and 35 years
* healthy at menacme, eutrophic, nulliparous
* functional evaluation of pelvic floor muscles presenting muscular strength ≥3 of the Oxford Scale.

Exclusion Criteria:

* Pregnant women will be excluded from the study;
* women with a history of previous abdominal and / or pelvic surgeries;
* urogynecological and neuromuscular diseases;
* vaginismus;
* increased perineal muscle tone;
* chronic constipation;
* diabetes;
* connective tissue disease;
* anal fissures;
* active hemorrhoids; (chronic pelvic pain, pyriform syndrome, hyperlordosis or marked lumbar rectification)
* smokers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activation of pelvic floor muscles | one day
  The electromyographic signal (RMS AEMFNPI) during the four pelvic patterns: anterior elevation, posterior elevation, anterior depression and posterior depression will be made as the lateral decubitus individual and in each muscle or muscle group evaluated during the execution of the combination technique isotonic in each pattern. The electromyographic recording of the abdominal and pelvic floor muscles will be done three times to perform the weighted average in the following sequences:
  Combination of isotonic (concentric, stabilizing and eccentric) of the anterior elevation pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the previous depression pattern; Combination of isotonic (concentric, stabilizing and eccentric) of the posterior elevation pattern;

SECONDARY OUTCOMES:
Motor learning after repetitive training of pelvic PNF patterns | 6 weeks
  The training of PNF pelvic patterns for motor learning in GI will be performed twice a week by a trained and experienced researcher for six weeks (CHRISTIANSEN et al., 2017). At each training session, there will be three repeated movements in each pelvic pattern.

OTHER OUTCOMES:
Body Mass Index (BMI) | one day
  weight and height will be combined to report BMI in Kg/m2
Sexual Function | one day
  ordinal qualitative variable, which will be measured through the Female Sexual Function Index (FSFI). Score 26 will be used as the cut-off point for categorizing the variable, in which scores ≤ 26 indicate sexual dysfunction.
Strength of pelvic floor muscles | one day
  a qualitative ordinal variable, which will be measured by the Oxford Scale, classified as: (0) Degree 0; (1) Grade 1; (2) Grade 2; (3) Grade 3; (4) Grade 4.
Postural change (pelvis) | one day
  continuous quantitative variable, measured through angulation in degrees during photogrammetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Josepha Karinne de Oliveira Ferro, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided